CLINICAL TRIAL: NCT02747030
Title: Phase I Study on the Feasibility and Safety of Surgical Stabilizer Assisted Retinal Vein Cannulation With Ocriplasmin Infusion for Central Retinal Vein Occlusion.
Brief Title: Phase I RVC With Ocriplasmin for CRVO
Acronym: RVC_CRVO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S58782
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2017-11

CONDITIONS: Central Retinal Vein Occlusion
Keywords: Central retinal vein occlusion; Retinal endovascular surgery; Retinal vein cannulation; Ocriplasmin
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Plasminogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ocriplasmin intravenously (Experimental): All subjects included in this phase I study are in the experimental treatment arm and will undergo a vitrectomy augmented with retinal vein cannulation and intravenous Ocriplasmin infusion.
  Interventions: Drug: Ocriplasmin intravenously

INTERVENTIONS:
Drug: Ocriplasmin intravenously — Retinal vein cannulation with Ocriplasmin infusion
  Other Names: Jetrea

SUMMARY:
In central retinal vein occlusion (CRVO) a blood clot blocks the venous outflow of the entire retinal circulation. This leads to retinal and vitreous hemorrhages, retinal edema and neovascularization. The development of a microneedle and surgical stabilizer made it possible to perform a prolonged (10 minutes) retinal vein cannulation with infusion of Ocriplasmin. Ocriplasmin has the advantage over tissue Plasminogen Activator (tPA) that it already is an active enzyme and a strong fibrinolyticum. This study aims to investigate the feasibility and safety of local intravenous Ocriplasmin for CRVO.

DETAILED DESCRIPTION:
Central retinal vein occlusion (CRVO) is the second most common source of permanent blindness in the Western world after diabetic retinopathy. By blocking the outflow pathway for the retinal circulation, visual prognosis is bad on the short and long term. Currently, treatment is mostly focused on treating the secondary effects: macular edema and neovascularization with antiVEGF and/or corticosteroid intravitreal injections and retinal laser photocoagulation. There is however a surgical treatment aimed at displacing the blood clot; a radial optic neurotomy. During this surgical treatment, the vitreous is removed by vitrectomy, after which a radial incision is made in the optic disc. The target of this incision is to open the canal in the lamina cribrosa to improve the blood flow in the central retinal vein. Since the outcome of this procedure is variable and has its inherent risks, mainly because the incision can damage the central retinal artery which is adjacent to the central vein, this procedure is not routinely performed in all vitreoretinal centers.

Following the recent development of a surgical stabilizer and microneedle suitable for retinal vein cannulations, the option for local intravenous administration of fibrinolytic drugs exists. This phase I study aims to investigate the feasibility and safety of surgical stabilizer assisted retinal vein cannulation with local intravenous infusion of Ocriplasmin to dissolve the clot clogging the central retinal vein. Ocriplasmin is the small active part of the larger plasmin molecule. Plasmin itself is formed by enzymatic conversion from plasminogen, a process that is mediated by tissue plasminogen activator (tPA). The amount of plasmin that can be produced is thus highly dependent on the amount of plasminogen that is present nearby the clot. By using Ocriplasmin, this intermediate step can be skipped and the clot will be targeted directly and during the entire time of infusion. By being able to get infusion times up to 10 minutes, abundant clot exposure to Ocriplasmin is guaranteed.

Inclusion will be offered to patients presenting with a recent CRVO, a vitrectomy will be performed augmented with retinal vein cannulation and infusion of ocriplasmin during 10 minutes.

Patients presenting with a recent CRVO (<2weeks) will be offered inclusion to undergo a vitrectomy with subsequent prolonged retinal vein cannulation and infusion of Ocirplasmin. The surgery is done by placing a microneedle in one of the branch retinal veins at the border of the optic disc. To increase the safety of this procedure a surgical stabilizer was developed. This procedure was abundantly tested and refined in multiple in vivo porcine experiments and the medication (Ocriplasmin) has already been tested for fibrinolytic activity used in 100-fold higher dosis intravenously and intra-arterially.

After the surgery, standard of care follow up with a comprehensive ophthalmological examination and technical investigations is foreseen. The primary outcome measures of this safety and feasiblity study are: technical success to cannulate the retinal vein and inject ocriplasmin to remove the blood clot, number of intervention-related (surgical or pharmacological) complications, duration of infusion.

If necessary; depending on the disease evolution, additional interventions like intravitreal antiVEGF, steroids or laser photocoagulation can be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Recent diagnosis of CRVO
* Onset of symptoms <10 days
* Visual acuity < 2/10 in study eye
* Visual acuity >1/10 in fellow eye
* Central macular thickness >250µm and <1000 µm
* Signed informed consent prior to inclusion

Exclusion Criteria:

* Fluorescein allergy
* Active neovascularization (NVD/NVE/NVI/NVA)
* Eye disease other than CRVO or Cataract decreasing vision
* Use of acetazolamide or other drugs potentially affecting macular edema, including systemic steroids >10mg/d
* History of retinal surgery
* High myopia (> -10D)
* Contraindication for the use of systemic anticoagulant medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12; Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Feasibility | peroperative
  technical succes of retinal vein cannulation and duration of infusion time
Safety | peroperative until 2 weeks postoperative
  number of intervention-related (surgical or pharmacological) complications

SECONDARY OUTCOMES:
central macular thickness | 2 weeks
  change in central macular thickness as measured with optical coherence tomography
surface of non-perfused retina | 2 weeks
  change in surface of non-perfused retina as measured with fluo-angiography
visual acuity | 2 weeks
  change in visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Overdam KA, Missotten T, Spielberg LH. Updated cannulation technique for tissue plasminogen activator injection into peripapillary retinal vein for central retinal vein occlusion. Acta Ophthalmol. 2015 Dec;93(8):739-44. doi: 10.1111/aos.12830. Epub 2015 Aug 27. PMID 26310993
- [Background] Verhamme P, Heye S, Peerlinck K, Cahillane G, Tangelder M, Fourneau I, Daenens K, Belmans A, Pakola S, Verhaeghe R, Maleux G. Catheter-directed thrombolysis with microplasmin for acute peripheral arterial occlusion (PAO): an exploratory study. Int Angiol. 2012 Jun;31(3):289-96. PMID 22634985
- [Background] Thijs VN, Peeters A, Vosko M, Aichner F, Schellinger PD, Schneider D, Neumann-Haefelin T, Rother J, Davalos A, Wahlgren N, Verhamme P. Randomized, placebo-controlled, dose-ranging clinical trial of intravenous microplasmin in patients with acute ischemic stroke. Stroke. 2009 Dec;40(12):3789-95. doi: 10.1161/STROKEAHA.109.560201. Epub 2009 Oct 15. PMID 19834019
- [Background] Verhamme P, Jerome M, Goossens G, Devis J, Maleux G, Stas M. A pilot trial of microplasmin in patients with long-term venous access catheter thrombosis. J Thromb Thrombolysis. 2009 Nov;28(4):477-81. doi: 10.1007/s11239-009-0310-x. Epub 2009 Feb 19. PMID 19225865